CLINICAL TRIAL: NCT01811056
Title: Exploring a Patient-centered Approach to Mifepristone Administration in Medical Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1006
Record Dates: First submitted 2013-03-11; First posted 2013-03-14 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Termination of Pregnancy
Keywords: medical abortion; mifepristone
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- In-Center Use of Mifepristone (No Intervention): Participants who choose to take mifepristone in the center
- Out-of-Center Use of Mifepristone (Experimental): Participants who choose to take the mifepristone outside of the center
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Mifepristone use outside of the center
  Other Names: mifeprex
  Arms: Out-of-Center Use of Mifepristone

SUMMARY:
This study will test ways to give women more options and flexibility when they are ending their unwanted pregnancies. The investigators will look at uptake and acceptability of using mifepristone outside of the clinic for pregnancy termination.

DETAILED DESCRIPTION:
This study will investigate the uptake of mifepristone administration outside of the health center for pregnancy termination and its acceptability to women and to their providers. In addition, we plan to evaluate rates of follow-up, adherence, efficacy, complications, days of missed work and/or school, and lost income. This will be a prospective, comparative, non-randomized, open-label study. All women who are seeking medical abortion will be offered participation in the study. Women who enroll in the study will be given a choice between taking the mifepristone outside the center or in the center setting.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years and older
* seeking medical abortion services
* in general good health
* assessed by a clinician to have an intrauterine pregnancy less than 64 days L.M.P on the day mifepristone will be taken
* eligible for medical abortion according to clinician and center standards.

Exclusion Criteria:

* will be followed up by beta HCG and not ultrasound

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2013-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who would choose outside of center administration of mifepristone again | 1-2 weeks
Proportion of participants who would recommend outside-of-center administration to a friend | 1-2 weeks

SECONDARY OUTCOMES:
Proportion of women who select outside-of-clinic use of mifepristone | 1-2 weeks
Success Rates/Method Failure | 1-2 weeks
  Ongoing pregnancy at study end Incomplete abortion at study end Medically indicated surgical intervention during study
Adherence | 1-2 weeks
  Did not take complete therapy Mifepristone not taken at scheduled time Mifepristone not taken within 63 days L.M.P. Misoprostol not taken within 48 hours of mifepristone administration Did not return for confirmation of outcome
Provider-related outcomes | 1-2 weeks
  Unscheduled visits to center Unscheduled calls to center/clinician on-call Provider satisfaction- better than center mifepristone, equivalent, or worse; impact on workload; impact on quality of care

OTHER OUTCOMES:
Productivity | 1-2 weeks
  Missed days of school and/or work Additional costs for childcare or eldercare
Reasons for selection of mifepristone administration site and experiences with home administration Reason | 1-2 weeks
  Reasons for selection of mifepristone administration site and experiences with home administration

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (3):
- United States (3):
  - Planned Parenthood of New York City, New York, New York
  - Planned Parenthood of Northern New England, Barre, Burlington, Rutland, Vermont
  - Planned Parenthood of the Great Northwest, Seattle, Washington

REFERENCES:
- [Background] Swica Y, Chong E, Middleton T, Prine L, Gold M, Schreiber CA, Winikoff B. Acceptability of home use of mifepristone for medical abortion. Contraception. 2013 Jul;88(1):122-7. doi: 10.1016/j.contraception.2012.10.021. Epub 2012 Nov 21. PMID 23177917
- [Result] Chong E, Frye LJ, Castle J, Dean G, Kuehl L, Winikoff B. A prospective, non-randomized study of home use of mifepristone for medical abortion in the U.S. Contraception. 2015 Sep;92(3):215-9. doi: 10.1016/j.contraception.2015.06.026. Epub 2015 Jul 2. PMID 26142620
- See also: Gynuity Health Projects Website — http://www.gynuity.org